CLINICAL TRIAL: NCT04196543
Title: Interest of a Post-operative Ultrasound With Systematic Use of Ultrasonic Contrast in the Follow-up of Aortic Endoprosthesis: Prospective Study at the University Hospital of Nice
Acronym: Ultra_Evar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-AOI-05
Record Dates: First submitted 2019-11-13; First posted 2019-12-12 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Aneurysm, Abdominal Aortic
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- écho-doppler with ultrasonar Sonovue® injection (Experimental)
  Interventions: Other: écho-doppler with ultrasonar Sonovue® injection

INTERVENTIONS:
Other: écho-doppler with ultrasonar Sonovue® injection — During this unique visit they will benefit from 2 imaging exams performed by two different operators:
  * Echo-doppler without "standard method" contrast injection (common practice)
  * An echo-doppler with Sonovue® ultrasound injection "Ultra_evar method" (2.5 ml bolus 2-3 seconds) During this examination, the endoprosthesis and the aneurysm sac will be scanned according to the 4 incidences described above in order to objective whether or not there is a endoleak.
  The patient then performs the control CT-scan prior to discharge from hospital.
  The results of the medical imaging exams will be communicated to them before the hospital discharge, once the CT-scan has been performed.
  A cross-review of the studies will be performed later.

SUMMARY:
This is a prospective study conducted on a population with an aortic endoprosthesis in the context of an abdominal aortic aneurysm. The study's objective is to standardize the ultrasound methodology in the monitoring of aortic endoprosthesis in immediate post-operative care by comparing the results with CT-scan (gold standard). To improve ultrasound methodology, the investigators propose to use the VESMA protocol for ultrasound diameter measurement at four incidences. In addition, the use of ultrasonic contrast agents increases the accuracy of vascular structures, the quality of the ultrasound blood flow image and the duration of signal enhancement. This makes it possible to visualize small gauge vessels and those with slow flows. In this way, the investigators could improve the ultrasound technique for measuring aneurysm bag diameters and endoleak detection. Moreover, the toxicity of iodinated contrast agents is the third cause of acute renal failure in hospitalized patients and is all the more frequent when the investigators increase injections. Improving the quality of ultrasound investigations for the monitoring of aortic endoprosthesis would therefore allow us to reduce the number of CT-scan performed in this population and thus reduce irradiation and the injection of nephrotoxic products. Thereby, the investigators would like to integrate the technique into the systematic follow-up of patients who have benefited from the placement of an aortic endoprosthesis by replacing the CT-scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Abdominal aortic aneurysm treated with aortic stent.
* Signature of informed consent.
* Person affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Hypersensitivity to sulphur hexafluoride or to these excipients (Macrogol 4000, Distearoylphosphatidylcholine, Dipalmitoylphosphatidylglycerol sodé, Palmitic acid).
* Right-left shunt patient
* Patient with severe pulmonary hypertension (pulmonary blood pressure > 90 mm Hg),
* Patient with uncontrolled systemic hypertension
* Adult patients with respiratory distress syndrome.
* Dobutamine patient in patients with a pathology suggesting cardiac instability
* Hypercoagulation, recent thromboembolic accident
* Fenestrated aortic stent
* Pregnant or nursing woman.
* Severe heart failure.
* Person deprived of liberty by judicial or administrative decision.
* Person subject to legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
measurement of anterior-posterior diameters according to 4 aortic endoprosthesis incidences after PCUS injection in immediate post-operative | 1 day
detection of endoleaks after PCUS injection in immediate post-operative | 1 day
measurement of anterior-posterior diameters of endoleaks after PCUS injection in immediate post-operative | 1 day

SECONDARY OUTCOMES:
Description of endoleaks after PCUS injection in immediate post-operative | 1 day
Description of exit doors of heart after PCUS injection in immediate post-operative | 1 day
Description of their flows after PCUS injection in immediate post-operative | 1 day
Description of maximum circulatory speeds after PCUS injection in immediate post-operative | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pascal GIORDANA, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- University Hospital of Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnston KW, Rutherford RB, Tilson MD, Shah DM, Hollier L, Stanley JC. Suggested standards for reporting on arterial aneurysms. Subcommittee on Reporting Standards for Arterial Aneurysms, Ad Hoc Committee on Reporting Standards, Society for Vascular Surgery and North American Chapter, International Society for Cardiovascular Surgery. J Vasc Surg. 1991 Mar;13(3):452-8. doi: 10.1067/mva.1991.26737. PMID 1999868
- [Background] Manning BJ, Kristmundsson T, Sonesson B, Resch T. Abdominal aortic aneurysm diameter: a comparison of ultrasound measurements with those from standard and three-dimensional computed tomography reconstruction. J Vasc Surg. 2009 Aug;50(2):263-8. doi: 10.1016/j.jvs.2009.02.243. PMID 19631858
- [Background] Bredahl KK. Response to commentary on "Re: Contrast Enhanced Ultrasound can Replace Computed Tomography Angiography for Surveillance After Endovascular Aortic Aneurysm Repair". Eur J Vasc Endovasc Surg. 2017 Mar;53(3):446-447. doi: 10.1016/j.ejvs.2016.12.029. Epub 2017 Jan 26. No abstract available. PMID 28131537